CLINICAL TRIAL: NCT05340621
Title: NAUTILUS: a Phase 1b/2 Study of OKI-179 Plus Binimetinib in Patients with Advanced Solid Tumors and Activating Mutations in the RAS Pathway (Phase 1b) and in Patients with Advanced NRAS-Mutated Melanoma (Phase 2)
Brief Title: NAUTILUS: OKI-179 Plus Binimetinib in Patients with Advanced Solid Tumors in the RAS Pathway (Phase 1b) and NRAS-mutated Melanoma (Phase 2)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OnKure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OKI-179-230
Record Dates: First submitted 2022-02-22; First posted 2022-04-22 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: RAS Mutation; NRAS Gene Mutation; Melanoma
MeSH Terms: conditions — Melanoma | interventions — binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- OKI-179 + binimetinib (Experimental)
  Interventions: Drug: OKI-179 + binimetinib

INTERVENTIONS:
Drug: OKI-179 + binimetinib — Phase 1b: With a 3+3 dose escalation design, enrollment in Phase 1b will proceed until the MTD has been defined or the highest dose level has been reached. OKI-179 will be administered on a 4-days-on/3-days-off schedule, while binimetinib will be administered BID continuously.
  Phase 2: Patients will be treated with the RP2D.

SUMMARY:
The NAUTILUS study is a Phase 1b/2, multi-center, open-label study in which patients with activating mutations in the RAS pathway (Phase 1b) and patients with NRAS-mutated Melanoma (Phase 2) will be treated with a combination of oral OKI-179 combined with the MEK inhibitor binimetinib.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1b: Solid tumor refractory to standard treatment, for which no standard therapy is available, or if the patient refuses standard therapy
* Phase 1b: Tumor has an activating mutation in the RAS pathway confirmed by any local or central laboratory, including but not limited to RAS, BRAF, NF1, and GNAQ/11
* Phase 1b: Prior MEK inhibitor exposure may be allowed per Sponsor agreement
* Phase 2: Histologically confirmed, metastatic melanoma with a confirmed NRAS mutation determined by a validated NRAS mutation detection kit performed in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory
* Phase 2: Prior ICI treatment with a programmed cell death 1 (PD-1) or programmed death ligand 1 (PD-L1) checkpoint inhibitor, or ineligible for this type of therapy
* Phase 2: Consent for a tumor biopsy or can provide a recent archival tumor biopsy sample (within 2 years)
* Phase 2: At least 1 measurable lesion based on RECIST version 1.1
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1.5 × 109/L
  * Platelets ≥ 100,000/μL
  * Hemoglobin ≥ 9.0 g/dL (at least 1 week after packed red blood cells, if applicable)
  * Total bilirubin within institutional ULN, unless patient has Gilbert's syndrome and has total bilirubin ≤ 2.5 × institutional ULN
  * Alanine aminotransferase and aspartate aminotransferase ≤ 2.5 × institutional ULN or < 5 × institutional ULN in the presence of liver metastasis
  * Serum creatinine < 1.5 × institutional ULN
* All prior treatment-related toxicities must have resolved to CTCAE version 5.0 criteria of Grade ≤ 1, except for alopecia and ICI-related endocrinopathies managed with hormone replacement therapy (eg, thyroiditis/hypothyroidism, hypophysitis, diabetes mellitus type 1)
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Able to swallow and tolerate oral medications
* Life expectancy ≥ 3 months

Exclusion Criteria:

* Any of the prior treatments, as described below:

  * Major surgery within 28 days of C1D1
  * Chemotherapy or radiation within 2 weeks of C1D1
  * Investigational agents within 4 weeks of C1D1 or < 5 half-lives, whichever is shorter, or expected toxicity not resolved to CTCAE version 5.0 criteria of Grade ≤ 1, except for alopecia and ICI-related endocrinopathies managed with hormone replacement therapy
  * Prior histone deacetylases inhibitors, MEK inhibitors (Phase 2 only), pan-deacetylating agents, or valproic acid for the treatment of cancer
  * Untreated or symptomatic brain metastasis. Patients with previously treated brain metastasis who are not on corticosteroids and are clinically stable are eligible for enrollment, as are patients with small (< 0.5 cm) untreated and asymptomatic brain metastases
* Known hypersensitivity to binimetinib or other MEK inhibitors
* Women who are pregnant or nursing
* Concomitant active malignancies or previous malignancies with < 2-year disease-free interval at the time of enrollment. Patients with adequately resected basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, stage 1 prostate cancer, or other malignancies deemed to be cured by prior therapy in the judgment of the Investigator may enroll irrespective of the time of diagnosis
* Any severe concurrent medical or psychiatric condition (including active systemic infection requiring intravenous antibiotics, uncontrolled diabetes mellitus, symptomatic congestive heart failure, uncontrolled hypertension, or cardiac arrhythmia) which, in the judgment of the Investigator, would make the patient inappropriate for study participation
* Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

  * History of acute myocardial infarction, acute coronary syndromes (including unstable angina, coronary artery bypass graft, coronary angioplasty or stenting) < 6 months prior to start of study treatment
  * Symptomatic congestive heart failure (Grade 2 or higher), history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality < 6 months prior to the start of study treatment, except medically managed atrial fibrillation or paroxysmal supraventricular tachycardia
  * Uncontrolled arterial hypertension despite medical management
* History or evidence of central serous retinopathy (CSR), retinal vein occlusion (RVO) or any eye condition that would be considered a risk factor for CSR or RVO, such as uncontrolled glaucoma or ocular hypertension
* Known previous or current serious ophthalmic disease, history of cataract surgery within < 8 days, serious eye trauma, or intraocular or ocular surgery other than refractive surgery (i.e. LASIK, cataract); patients with uveal melanoma/eye enucleation due to uveal melanoma are permitted to enroll
* Patients who have neuromuscular disorders that are associated with elevated creatine phosphokinase (CPK; eg, inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy) or elevated baseline CPK levels (≥ Grade 2)
* History of recent (≤ 90 days) thromboembolic or cerebrovascular event such as transient ischemic attack, cerebrovascular accident, or hemodynamically significant (massive or submassive) deep vein thrombosis or pulmonary emboli (DVT/PE). Note: Patients with DVT/PE that does not result in hemodynamic instability may enroll as long as they are anticoagulated for at least 4 weeks. Note: Patients with DVT/PE related to indwelling catheters or other procedures may enroll
* Any medical condition that would impair the administration of oral agents, such as active inflammatory bowel disease or uncontrolled nausea, vomiting, or diarrhea
* Known positive serology for HIV and AIDS-related illness with CD4 count < 350/mL and/or known active hepatitis B or hepatitis C. Testing prior to C1D1 is not required
* History or current evidence of congenital long QT syndrome
* QTcF corrected with Fridericia's formula > 470 msec on screening electrocardiogram (ECG)
* Ongoing medication that leads to significant QT prolongation
* Ongoing medication that is a strong cytochrome P450 3A4 inhibitor or inducer
* Ongoing medication that is a strong inhibitor of P-glycoprotein and sensitive substrates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Phase 1b: Incidence and severity of dose-limiting toxicities (DLTs) | First 28 days of treatment
  Incidence and severity of DLTs will be measured in the DLT-evaluable population during Cycle 1.
Phase 1b: Incidence and severity of adverse events (AEs) | Phase 1b study duration (approximately 1.5 years)
  AEs will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Phase 1b: Change in clinical laboratory abnormalities | Baseline through 30 days after end of study treatment
  Changes from baseline through study treatment will be analyzed using NCI CTCAE version 5.0 grade criteria
Phase 1b: Change in Eastern Cooperative Oncology Group (ECOG) performance status | Phase 1b study duration (approximately 1.5 years)
Phase 2: Objective response rate (ORR) | Phase 2 study duration (approximately 3 years)
  Objective responses will be determined per RECIST version 1.1 criteria, and the ORR will be defined as the proportion of patients with the best overall confirmed response of complete response (CR) or partial response (PR) in the Efficacy-Evaluable Population

SECONDARY OUTCOMES:
Phase 1b: Peak plasma concentration (Cmax) of OKI-179 and OKI-006 | First 28 days of treatment
  PK parameters will be measured based on plasma concentration-time data of OKI-179 and OKI-006
Phase 1b: Area Under the Plasma Concentration vs. Time Curve (AUC) of OKI-179 and OKI-006 | First 28 days of treatment
  PK parameters will be measured based on plasma concentration-time data of OKI-179 and OKI-006
Phase 1b: Objective response rate (ORR) | Phase 1b study duration (approximately 1.5 years)
  Objective responses will be determined per RECIST version 1.1 criteria, and the ORR will be defined as the proportion of patients with the best overall confirmed response of complete response (CR) or partial response (PR) in the Efficacy-Evaluable Population.
Phase 1b: Clinical Benefit Rate (CBR) | Phase 1b study duration (approximately 1.5 years)
  Clinical benefit will be defined as the best overall confirmed response of CR, PR or stable disease for at least 3 months. The CBR will be defined as the proportion of patients with clinical benefit in the Efficacy-Evaluable Population.
Phase 1b: Duration of Response (DOR) | Phase 1b study duration (approximately 1.5 years)
  The DOR will be calculated for all patients achieving a confirmed CR or PR and will be defined as the time from first disease assessment of PR or CR (whichever is first recorded) to the end of response, defined as occurrence of PD, death due to any cause, or relapse from CR.
Phase 2: Peak plasma concentration (Cmax) of OKI-179 and OKI-006 | First 28 days of treatment
  PK parameters will be measured based on plasma concentration-time data of OKI-179 and OKI-006
Phase 2: Area Under the Plasma Concentration vs. Time Curve (AUC) of OKI-179 and OKI-006 | First 28 days of treatment
  PK parameters will be measured based on plasma concentration-time data of OKI-179 and OKI-006
Phase 2: Progression-free survival (PFS) | Phase 2 study duration (approximately 3 years)
  Progression-free survival will be defined as the time from the first administration of OKI-179 to the date of progression or death due to any cause.
Phase 2: Clinical Benefit Rate | Phase 2 study duration (approximately 3 years)
  Clinical benefit will be defined as the best overall confirmed response of CR, PR or stable disease for at least 3 months. The CBR will be defined as the proportion of patients with clinical benefit in the Efficacy-Evaluable Population.
Phase 2: Duration of Response | Phase 2 study duration (approximately 3 years)
  The DOR will be calculated for all patients achieving a confirmed CR or PR and will be defined as the time from first disease assessment of PR or CR (whichever is first recorded) to the end of response, defined as occurrence of PD, death due to any cause, or relapse from CR.
Phase 2: Incidence and severity of AEs | Phase 2 study duration (approximately 3 years)
  AEs will be graded according to the NCI CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Sullivan, MD, Principal Investigator — Massachusetts General Hospital
Locations (12):
- United States (12):
  - CTCA Phoenix, part of City of Hope, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California
  - University of Florida Health Cancer Center, Gainesville, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - CTCA Atlanta, part of City of Hope, Newnan, Georgia
  - CTCA Chicago, part of City of Hope, Zion, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No